CLINICAL TRIAL: NCT00061919
Title: A Phase III Randomized, Double Blind, Placebo Controlled Trial Of Carboplatin/Etoposide With Or Without Thalidomide In Small Cell Lung Cancer (Study 12)
Brief Title: Carboplatin and Etoposide With or Without Thalidomide in Treating Patients With Limited-Stage or Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000302440; LLCG-STUDY-12 (Other: UCL CTC); EU-20207 (Other: UCL CTC); ISRCTN16174527 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Etoposide; Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active arm (thalidomide) (Experimental): Carboplatin IV on day 1 and etoposide IV on day 1 and 2 and, orally Day 3. Oral thalidomide daily beginning on day 1 for up to 24 months.
  Interventions: Drug: Carboplatin, etoposide & thalidomide
- Placebo arm (Placebo Comparator): Carboplatin IV on day 1 and etoposide IV on day 1 and 2 and, orally Day 3. Oral placebo daily beginning on day 1 for up to 24 months.
  Interventions: Drug: Carboplatin, etoposide & placebo

INTERVENTIONS:
Drug: Carboplatin, etoposide & thalidomide — Carboplatin IV on day 1 and etoposide IV on day 1 and 2 and, orally Day 3. Oral thalidomide daily beginning on day 1 for up to 24 months.
  Arms: Active arm (thalidomide)
Drug: Carboplatin, etoposide & placebo — Carboplatin IV on day 1 and etoposide IV on day 1 and 2 and, orally Day 3. Oral placebo daily beginning on day 1 for up to 24 months.
  Arms: Placebo arm

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as carboplatin and etoposide use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. It is not yet known if combination chemotherapy is more effective with or without thalidomide in treating small cell lung cancer.

PURPOSE: This randomized phase III trial is studying carboplatin, etoposide, and thalidomide to see how well they work compared to carboplatin and etoposide in treating patients with limited- or extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with limited or extensive stage small cell lung cancer treated with carboplatin and etoposide with vs without thalidomide.
* Compare the time to disease progression in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the response rates of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease stage (limited vs extensive), ECOG performance status (0 and 1 vs 2), and alkaline phosphatase (no greater than 1.5 times upper limit of normal [ULN] vs greater than 1.5 times ULN). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carboplatin IV over 30 minutes on day 1 and etoposide* IV over 1-2 hours on days 1 and 2 and orally on day 3. Patients also receive oral thalidomide daily beginning on day 1.
* Arm II: Patients receive carboplatin and etoposide as in arm I and oral placebo daily beginning on day 1.

NOTE: *Patients who are unable to receive etoposide IV on day 2 may receive oral etoposide on days 2 and 3.

In both arms, chemotherapy (carboplatin and etoposide) repeats every 3 weeks for up to 6 courses. Patients receive thalidomide or placebo continuously for up to 2 years. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may continue to receive thalidomide or placebo provided the patient is clinically and symptomatically stable.

Quality of life is assessed at baseline, during each course of chemotherapy, at 3-4 weeks after completion of chemotherapy, and at 6, 12, 18, and 24 months.

Patients are followed every 2 months for 2 years after the completion of chemotherapy and then every 3 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 372 patients (186 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Limited or extensive stage disease
* No symptomatic brain metastases requiring immediate radiotherapy

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-3

Life expectancy

* At least 8 weeks

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Ethylenediamine tetraacetic acid (EDTA) clearance greater than 60 mL/min OR
* Creatinine clearance greater than 50 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception (including 1 highly effective method and 1 barrier method) during and for 4 weeks after study completion
* No other prior malignancy within the past 3 years except nonmelanoma skin cancer or early cervical cancer
* No significant medical condition or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2003-04; Primary Completion 2007-02 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Survival at 2 years after study randomization | 0-2 years

SECONDARY OUTCOMES:
Time to disease progression 2 years after study randomization | 0-2 years
Toxicity as measured by NCIC CTC 3 times weekly while undergoing chemotherapy, then monthly thereafter | Till end of treatment
Response rates as measured by RECIST during each visit while undergoing chemotherapy and after completion of study treatment | Till progression
Quality of life as measured by EORTC QLQ-30 and lung-specific questionnaire(LC14) at baseline, after each course, and after completion of study treatment, and at 6, 12, 18, and 24 months after day 1 of course 1 | 0-24 months
Biological markers (measurement of VEGF, bFGF, TNF alpha, and IL-6) | Before treatment courses 1 and 4, and then at 9 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Siow M. Lee, MD, PhD, FRCP, Study Chair — University College London Hospitals
Locations (1):
- University College of London Hospitals, London, England, United Kingdom

REFERENCES:
- [Result] Lee SM, Woll PJ, Rudd R, Ferry D, O'Brien M, Middleton G, Spiro S, James L, Ali K, Jitlal M, Hackshaw A. Anti-angiogenic therapy using thalidomide combined with chemotherapy in small cell lung cancer: a randomized, double-blind, placebo-controlled trial. J Natl Cancer Inst. 2009 Aug 5;101(15):1049-57. doi: 10.1093/jnci/djp200. Epub 2009 Jul 16. PMID 19608997